CLINICAL TRIAL: NCT01376102
Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance to Monitor the Safety of BONVIVA(Ibandronate) Injection Administered in Korean Patients According to the Prescribing Information
Brief Title: BONVIVA(Ibandronate) Injection PMS(Post-marketing Surveillance)
Acronym: BONINJPMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111412
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Osteoporosis
Keywords: osteoporosis; ibandronate
MeSH Terms: conditions — Osteoporosis | interventions — Injections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BONVIVA(ibandronate): Patients administrated ibandronate injection with postmenopausal osteoporosis
  Interventions: Drug: BONVIVA(ibandronate) injection

INTERVENTIONS:
Drug: BONVIVA(ibandronate) injection — Basically there is no treatment allocation. Subjects who would be administered of ibandronate at their physicians' discretion will be enrolled. Dosage regimen will be recommended according to the prescribing information. Subjects will be enrolled consecutively.

SUMMARY:
This is an open label, multi-centre, non-interventional post-marketing surveillance

DETAILED DESCRIPTION:
This is an open label, multi-centre, non-interventional post-marketing surveillance to monitor the safety of Ibandronate injection administered in postmenopausal osteoporosis patients according to the prescribing information

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at study entry:

Subjects administered with BONVIVA(ibandronate) injection following the locally approved prescribing information Women diagnosed with postmenopausal osteoporosis. Subjects who the investigator believes that they can and will comply with the requirements of the protocol Subjects with no experience of treatment using ibandronate injection Note: Subjects, who have experience of other bisphosphonates treatment, can be included.

Subjects who are indicated and administered of ibandronate injection according to the Prescribing Information in normal prescription use

Exclusion Criteria:

Considering the nature of this non-interventional PMS, there is no strict exclusion criteria set up. The doctors participating this study to enrol the subjects prescribed with ibandronate injection following the locally approved Prescribing Information.

The following criteria should be checked at the time of study entry.

According to contraindication on the prescribing information, ibandronate injection should not be administered to the following patients:

Patients with known hypersensitivity to ibandronate injection or to any of its excipients Uncorrected hypocalcemia Note: Ibandronate injection is not recommended for use in patients who have a serum creatinine above 200 μmol/l (2.3 mg/dl) or who have a creatinine clearance (measured or estimated) below 30 ml/min, because of limited clinical data available from studies including such patients.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients administrated BONVIVA(ibandronate) injection with postmenopausal osteoporosis
Sampling Method: Probability Sample
Enrollment: 657 (Actual)
Dates: Start 2007-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The number of adverse event after ibandronate administration | 6 months

SECONDARY OUTCOMES:
The number of unexpected adverse drug reaction after BONVIVA(ibandronate) injection administration | 6 months
The number of serious adverse event after BONVIVA(ibandronate) injection administration | 6 months
Effectiveness of BONVIVA(ibandronate) injection treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea